CLINICAL TRIAL: NCT00189072
Title: Effects of Pain and the Treatment of Pain With Gabapentin (900-3600 Mg) on Driving Ability, Attentional Capacity and Psychomotor Performance in Chronic Neuropathic Pain Patients
Brief Title: Effects of Gabapentin in the Treatment of Neuropathic Pain on Driving Performance and Cognition
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Utrecht University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 02/327
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2005-09-16 (Estimated); Status verified 2005-05

CONDITIONS: Chronic Neuropathic Pain
Keywords: gabapentin; neuropathic pain; driving; attention
MeSH Terms: conditions — Neuralgia | interventions — Gabapentin

INTERVENTIONS:
Drug: gabapentin

SUMMARY:
The aim of this study was to explore the effects of pain on the one hand and the effects of treatment of pain with gabapentin (900, 1200, 1800 or 2400 mg) on the other hand on actual driving performance and several laboratory tests in patients with neuropathic pain. It was hypothesized that gabapentin might influence performance after acute but not after subchronic administration.

DETAILED DESCRIPTION:
Numerous studies demonstrate neuropsychological impairment in patients with chronic pain, particularely on measures assessing attentional capacity, processing speed and psychomotor speed. About 50% of the patients suffering from neuropathic pain are treated with anticonvulsants, as a treatment against serious pain complaints, and experience good pain relief. Gabapentin is one of the most prescribed anticonvulsants for the treatment of neuropathic pain. An important disadvantage of treatment with gabapentin could be the occurrence of side effects, such as somnolence and fatigue. These side effects can constitute a crucial problem for patients treated with gabapentin who must operate a motor vehicle or other dangerous machinery. However, pain affects cognition negatively, and possibly also driving. Therefore, another possibility is that treatment with gabapentin for these pain complaints can improve driving because the pain has less influence. Since driving is an activity of daily living that is important in maintaining independency in the community, such as access to employment and social activities, it is important to establish the effects of using gabapentin on these abilities. No studies have been conducted so far to investigate driving abilities of patients with neuropathic pain, treated with gabapentin.The aim of this study was to explore the effects of pain on the one hand and the effects of acute (Day 1) and subchronic (Day 15) treatment of pain with gabapentin (900, 1200, 1800 or 2400 mg) on the other hand on actual driving performance and several laboratory tests in patients with neuropathic pain. It was hypothesized that gabapentin might influence performance after acute but not after subchronic administration. This study is a two-period double-blind, placebo-controlled, cross-over randomised study.

ELIGIBILITY:
Inclusion Criteria:

* age, responder to gabapentin,succesfully treated with gabapentin at least 4 weeks before start of study, minimal VAS pain intensity scores of 4 cm on a 10 cm scale, driving licence, driving experience, fluently speaking Dutch, normal vision, right-handed

Exclusion Criteria:

* alcohol- or drug dependence, use of other psychotropic medication, use of illicit drugs, psychological or physical disorder other than pain or pain-related, excessive smoking and drinking

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24
Dates: Start 2003-04

PRIMARY OUTCOMES:
driving test parameters

SECONDARY OUTCOMES:
laboratory test parameters
Event Related Potentials

CONTACTS AND LOCATIONS:
Overall Officials: Edmund Volkerts, PhD, Principal Investigator — Utrecht University
Locations (1):
- University of Utrecht, Utrecht, Utrecht, Netherlands